CLINICAL TRIAL: NCT03361215
Title: Disease Trajectories in Atopic Dermatitis and Psoriasis
Brief Title: Disease Trajectories and Anti-cytokine Response Signatures in Atopic Dermatitis and Psoriasis
Acronym: DiTrAP
Status: Recruiting | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stephan Weidinger, Prof. Dr. med., University Hospital Schleswig-Holstein
Other Study IDs: A100/12a1
Record Dates: First submitted 2017-11-27; First posted 2017-12-04 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis; Psoriasis; Healthy
Keywords: Disease progression; Disease course; Immunological characterization
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis; Disease Progression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, including EDTA, PBMC and serum samples for genetic and gene expression analysis Lesional and nonlesional biopsies (4 mm punch biopsies) for gene expression analysis Skin swabs for microbiome assessments Tape strips for protein analyis Stool samples for microbiome analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atopic dermatitis: Patients with dermatologist-diagnosed atopic dermatitis, psoriasis or autoimmune skin disease.
  Interventions: Other: Biosampling for molecular analysis
- Controls: Healthy volunteers with no history of atopic, autoimmune or chronic inflammatory disease.
  Interventions: Other: Biosampling for molecular analysis

INTERVENTIONS:
Other: Biosampling for molecular analysis — Observational study with no therapeutic intervention. Biosampling for molecular analysis

SUMMARY:
The clinical study investigates the long-term course of disease in patients with chronic inflammatory skin diseases (atopic eczema and psoriasis) and the impact of tarheted therapies on the clinical and molecular level. For this purpose, patients are asked to take part in regular examinations and data collections, and to donate biomaterials (blood, skin biopsies, skin swabs, tape strips, stool samples). Blood samples are used to analyze inflammation messengers. Punch biopsies from lesional and non-lesional skin areas are used to analyze gene expression. Tape strips are pieces of transparent adhesive tapes to strip off most of the horny layer that will be used to examine mRNA and protein expression. The skin smears are superficial smears of three areas of skin with cotton swabs, which are used to examine bacteria on the skin. Overall, the study will help to monitor the disease course clinically and on the molecular level in participating patients for at least ten years and to collect information about the impact of various external factors including treatments. The study has no effect on the therapies of the disease, it serves only the accompanying data collection

DETAILED DESCRIPTION:
Atopic dermatitis and psoriasis are the most common chronic inflammatory skin diseases in dermatology. Due to genetic predispositions, inflammatory changes of the skin occur. The specific mechanisms are only partly understood for both diseases and targeted therapies are established in psoriasis therapy and are becoming available for atopic dermatitis. In order to better understand the course of the disease and to characterize the changes in the inflammatory mechanisms during the course of the disease and under the influence of external factors such as therapies, longitudinal prospective studies are needed to evaluate clinical data and biological samples. This study investigates long-term clinical and epidemiological data from affected patients, as well as biological samples, including blood samples, skin biopsies, non-invasive skin swabs for microbiome detection, and tape strips for the molecular characterization of the disease. Data collection and biosampling will be done during routine visits, typically at week 0, 2, 4, 12 and 52.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of atopic dermatitis, psoriasis or autoimmune skin disease
* Written informed consent obtained from the subject

Exclusion Criteria:

* Patients who decline participation

In patients<18 years of age no biopsies will be taken

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient who are beeing treated in the routine care with chronic inflammatory skin diseases will be asked to participate in this project.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-03-16 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease progression | 10 years
  Epidemiological and phenotypical data of patients
Molecular signature changes | 10 years
  Molecular signatures will be measured using OMICS and sequencing technologies

SECONDARY OUTCOMES:
Development of comorbidities | 10 years
  Assessment of newly developed comorbid diseases over time

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Weidinger, Prof. Dr., Principal Investigator — Dept. of Dermatology University Hospital Kiel
Locations (1):
- Department of Dermatology, University Hospital Schleswig Holstein, Campus Kiel, Kiel, Germany